CLINICAL TRIAL: NCT01023607
Title: Evaluation of Statin-induced Lipid-rich Plaque Progression by Optical Coherence Tomography (OCT)Combined With Intravascular Ultrasound (IVUS)
Brief Title: Evaluation of Statin-induced Lipid-rich Plaque Progression by Optical Coherence Tomography (OCT) Combined With Intravascular Ultrasound (IVUS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yu Bo, Bo Yu ,President, Department of Cardiology, Harbin Medical University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HMUOCT-STATIN
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Coronary Artery Disease; Hyperlipidemia
Keywords: optical coherence tomography; intravascular ultrasound; Coronary artery disease; Hyperlipidemia
MeSH Terms: conditions — Coronary Artery Disease; Hyperlipidemias | interventions — Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A: (Active Comparator): Atorvastatin 20mg
  Interventions: Drug: Atorvastatin
- Group B: (Experimental): Atorvastatin 60mg
  Interventions: Drug: Atorvastatin
- Group C: (Active Comparator): Rosuvastatin 10mg
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 20mg/day
  Arms: Group A:
Drug: Atorvastatin — Atorvastatin, 60mg/day
  Arms: Group B:
Drug: Rosuvastatin — Rosuvastatin,10mg/day
  Arms: Group C:

SUMMARY:
Many trials suggested that lipid lowering therapy could significantly reduce cardiovascular events. Enhancing stability of vulnerable plaque is probably the main reason by which statins reduce adverse coronary events. The size of lipid core and the fibrous cap thickness (FCT) are the major determinants of plaque vulnerability. So, it is very important to accurately evaluate changes in plaque after stains therapy.

Previous reports suggested that intensive lipid lowering therapy provide more significantly clinical benefit compared with moderate lipid lowering therapy.Such benefit may contribute to the changes in following parameters: FCT, lipid arc(quadrants), TCFA, macrophage, plaque disruption, and thrombus measured by OCT, and plaque burden and remodeling index by IVUS.

Current intravascular imaging modalities, such as optical coherence tomography (OCT) and intravascular ultrasound (IVUS) can provide in vivo quantitative and qualitative information of coronary plaques. However, there were few studies aimed at monitoring the progression of coronary plaques in patients receiving statin therapy by OCT combined with IVUS.

Therefore, the study we designed were to compare the effect of the rosuvastatin 10mg, atorvastatin 20mg and atorvastatin 60mg treatment on the changes in FCT and lipid core arc by OCT and plaque burden by IVUS of coronary atherosclerotic plaques.

ELIGIBILITY:
Inclusion Criteria:

1. Age :18-75Y
2. Clinical indication for coronary angiography (CAG).
3. CAG demonstrates at least 1 de novo lesion with luminal diameter stenosis between 20% and 70% (visual estimation).
4. OCT demonstrates the lesion is a lipid-rich plaque (FCT ≤200μm and lipid arc ≥100o).
5. LDL-C range between 70mg /dl and 160mg /dl.
6. Patient or legal guardian understands and agrees to comply with all specified study requirements and provides written informed consent.

Exclusion criteria:

1. Life expectancy <12 months due to another medical condition.
2. Contraindication to the atorvastatin and rosuvastatin.
3. Creatinine levels more than 2.0mg/dL or ESRD.
4. Severe hepatic dysfunction (AST and/or ALT more than 3 times the upper limit of normal).
5. Congestive heart failure (left ventricle eject fraction ≤35%).
6. Female of childbearing potential with a positive pregnancy test within 7 days before study, or lactating, or intends to become pregnant during the following 12 months.
7. The patient is likely to require coronary bypass surgery, cardiac transplantation, surgical repair or replacement during the course.

Exit criteria

1. ALT/AST ≥ 3times upper limit of normal after enrollment.
2. Muscle ache/myopathy.
3. Lose follow-up.
4. Patient insists on exit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To compare the effects of atorvastatin 20mg and atorvastatin 60mg on the changes of FCT assessed by OCT and plaque burden by IVUS. | 12 months after enrollment

SECONDARY OUTCOMES:
To investigate the changes of FCT assessed by OCT and plaque burden by IVUS in comparisons of atorvastatin 60 mg vs rosuvastatin 10 mg, and atorvastatin 20 mg vs rosuvastatin 10 mg. | 12 months
To investigate the changes of remodeling index assessed by IVUS in comparisons of atorvastatin 60 mg vs atorvastatin 20 mg,atorvastatin 60 mg vs rosuvastatin 10 mg, and atorvastatin 20 mg vs rosuvastatin 10 mg | 12 months
To investigate the changes of macrophage infiltration semi-quantitatively by OCT in comparisons of atorvastatin 60 mg vs atorvastatin 20 mg,atorvastatin 60 mg vs rosuvastatin 10 mg, and atorvastatin 20 mg vs rosuvastatin 10 mg | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, MD,PhD, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (1):
- The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

REFERENCES:
- [Derived] Dong N, Xie Z, Wang W, Dai J, Sun M, Pu Z, Tian J, Yu B. Comparison of coronary arterial lumen dimensions on angiography and plaque characteristics on optical coherence tomography images and their changes induced by statin. BMC Med Imaging. 2016 Nov 22;16(1):63. doi: 10.1186/s12880-016-0166-4. PMID 27871242